CLINICAL TRIAL: NCT03655600
Title: Acupressure for Preventing Post-Operative Pain and Opioid Use Among Breast Cancer Patients Receiving Surgery
Brief Title: Acupressure for Pain and Opioid Use Among Breast Cancer Patients
Acronym: AcuPOP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting and retaining participants
Sponsor: University of Michigan (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency); Michigan Opioid Prescribing Engagement Network (Michigan-OPEN) (Unknown)
Responsible Party: Principal Investigator, Suzanna Zick, Assistant Research Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HUM00140468
Record Dates: First submitted 2018-08-06; First posted 2018-08-31 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer; Fatigue; Chronic Pain
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomized two arm (intervention and usual care) clinical trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-administered acupressure (Active Comparator): Acupressure administered by participant self-taught from computer application
  Interventions: Other: Self-administered acupressure
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Other: Self-administered acupressure — Self-administered acupressure learned through app for reduction of need for opioids post-surgery in breast cancer patients
  Arms: Self-administered acupressure

SUMMARY:
This study seeks to determine the feasibility of recruiting and training participants in self-acupressure, for women undergoing primary breast cancer surgery or delayed reconstruction surgery. The study seeks to determine also if self-acupressure is effective in reducing the need for opioids post-surgery and the effects on other life factors.

DETAILED DESCRIPTION:
Chronic pain following breast cancer surgery is a significant problem for women. There are over 3 million women in the United States living as breast cancer survivors. Sustained post-surgical pain is one of the most troubling side-effects for these women and continues to affect around 25-60% of breast cancer survivors, with approximately half classifying pain as being moderate to severe. Chronic cancer-related pain is associated with increased fatigue, depression, anxiety, sleep disruption, and decreased quality of life and function.

Acute pre- and post-operative pain are significant predictors of sustained pain following breast cancer surgery, but are insufficiently managed. The etiology of persistent breast cancer related pain following surgery is multifactorial and may be the direct effect of cancer or cancer treatment (e.g. surgery). Known risk factors for this chronic pain include younger age, higher body mass index, type of surgery (axillary lymph node dissection), and presence of a mood disturbance. Cancer patients may develop pain from neurotoxicity from adjuvant chemotherapy, and radiation may also play a role, and causes persistent pain in 13 - 26% of patients.

Two of the most significant factors that determine persistent pain following breast cancer surgery are the degree of pre-surgical pain and acute post-surgical pain. Recent reports have suggested that treatments aimed at reducing these factors may be effective at preventing the development of chronic pain following breast cancer surgery. Existing pre-emptive treatments to reduce this acute surgical pain include the use of nerve blocks and/or pharmacologic agents such as opioids, NSAIDs, ketamine, and gabapentin. While some pharmacologic approaches yield clinically meaningful reductions in post-operative pain in the research setting, there remains controversy in the field. For example in breast surgery specifically, a recent meta-analysis showed that thoracic paravertebral blocks have a statistically significant effect on reducing chronic pain, but the effect was not clinically meaningful and was associated with procedural risks such as vascular puncture.

In addition to the risk of developing pain following breast cancer surgery, women also report increased acute and chronic surgical pain following breast reconstruction surgery. In one of the first studies to examine pain post-reconstruction surgery, Wallace et al. found that the incidence of pain one year following breast cancer mastectomy plus reconstruction was 49% as compared to 31% for mastectomy alone. This increase was both statistically and clinically significant, and remains a current undertreated problem. Overall many women develop persistent pain after breast cancer surgery following either tumor removal or breast reconstruction. We know that this is influenced by acute pre- and post-surgical pain, but unfortunately the existing measures available for clinicians to prevent persistent post-surgical pain are not adequate.

Opioids are commonly used analgesics in the perioperative surgical setting; however, they are accompanied by significant limitations. Opioids are the most common pharmacologic intervention used for acute perioperative surgical pain. They are known to decrease pain via activation of specific receptors (mu, delta, and kappa), which inhibit neuronal firing resulting in reduced nociceptive activity. Although widely prescribed there are significant limitations for opioid use including tolerance, addiction, diversion, and even mortality. There were over 33,000 opioid deaths in the US in 2016 alone and the majority of these have been from opioid prescriptions. The US is currently experiencing an opioid epidemic wherein Americans constitute only 5% of the global population yet we consume over 80% of the world's opioid supply. Unfortunately, while opioids are needed in the surgical setting, the problem of increased opioid use is itself compounded by surgery. Patients receiving even low-risk surgeries are 44% more likely to become de novo long-term opioid consumers. With respect to breast cancer surgery, the odds of developing chronic opioid consumption following mastectomy increases by approximately 300%. Although the reason(s) for developing chronic opioid consumption are largely unknown, patients that receive a new opioid prescription within 7 days post-surgery, as compared to those who do not, are more likely to still be receiving opioids one year out. Thus acute pre-surgical and post-surgical pain, in addition to being risk factors for persistent chronic pain, may also increase the probability of becoming a chronic opioid consumer. There is an unmet need for analgesic interventions that are opioid sparing in the breast cancer surgical setting. This study proposes that acupressure may be one such option.

Acupressure Self-administered acupressure is one possible safe, self-management technique which may be effective for improving post-operative pain and opioid consumption. Acupressure, a technique derived from acupuncture, is a component of Traditional Chinese Medicine (TCM) in which pressure is applied to specific acupoints on the body using a finger or small device, to treat disease. Prior research has demonstrated that acupressure, self-administered by women with breast cancer, significantly reduced clinically significant pain by approximately one-third and was superior to standard therapies. Moreover, these self-rated improvements were maintained up to one month after treatment was discontinued.

Acupressure has been found to be effective for acute post-surgical pain, but no studies have examined the impact on the development of chronic pain or acute and chronic opioid use in any patient population. Four previous studies in diverse patient populations (appendectomy, cesarean section, gastric cancer, and knee arthroscopy) have found that acupressure delivered by an acupressure practitioner was able to significantly decrease post-surgical pain compared to either usual care or sham acupressure from as early as 60 minutes after surgery to as long as 3 days post-surgery, however no study has measured pain beyond 3 days post-surgery.29-32 As such, it is unknown what impact if any acupressure has on the development of chronic pain post-surgery. Also, no study has examined the impact of acupressure on either acute or chronic opioid use. In contrast, the one study that used an acuband (a band worn around the wrist with a nub over the acupressure point to provide stimulation) at the P6 point commonly used to treat nausea and vomiting had no impact on post-surgical pain 24 hours after receiving an appendectomy.

Along with a lack of research on acupressure's impact on chronic pain and opioid use the impact of this intervention on breast cancer patients undergoing surgery (mastectomy, lumpectomy, delayed or immediate reconstruction) is unknown. This study is a pilot randomized clinical trial to explore this intervention in 72 breast cancer patients scheduled for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of breast cancer stage 0 to III;
2. Planned unilateral or bilateral mastectomy or planned delayed breast reconstruction surgery within 24 months following unilateral or bilateral mastectomy;
3. For delayed breast reconstruction patients only: apparently cancer free at time of delayed reconstruction;
4. No planned new interventions for pain the two weeks prior to surgery;
5. Able to self-administer treatment at the specified points.

Exclusion Criteria:

1. Medically unstable (e.g. uncontrolled diabetes, high blood pressure, etc.);
2. For delayed breast reconstruction only: taking aromatase inhibitors which could confound surgical and chronic pain measurements;
3. Have a diagnosis of untreated mood disorder, e.g., bipolar or major depressive disorder;
4. Unwilling to maintain stable does of allowed chronic pain medications (e.g. NSAIDS, benzodiazepines, SSRIs and SNRIs);
5. Pregnant, those planning a pregnancy, or lactating mothers;
6. Any medical condition or treatment factor that the study team feels would either compromise the data acquired or introduce a potential safety concern.
7. Unable to give consent;
8. Acupuncture or acupressure receipt in past year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological females only
Enrollment: 8 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment for self-acupressure: Measure screening to on-study ratio of participants | 14 days
  Measure screening to on-study ratio of participants from Screening to Baseline
Feasibility of training, as measured by number of participants who complete the daily self-reported logbook | 28 days
  Measure the compliance of self-acupressure participants who are using the training application via daily self-reported logbook
Feasibility of training for self-acupressure: Measure the fidelity (accuracy) of participants using training application via instrument administered by study team | 1 day
  Measure the fidelity (accuracy) of participants using training application via instrument administered by study team

SECONDARY OUTCOMES:
Pain mitigation in acute postoperative period measured using the Brief Pain Inventory | 2 weeks
  Pain will be measured using the Brief Pain Inventory (0 being no pain and 10 being bad as can imagine)
Opioid use mitigation in acute postoperative period | 2 weeks
  Opioid use will be measured across both arms using oral morphine equivalents (OME)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna M Zick, ND, MPH, Principal Investigator — University of Michigan; Richard E Harris, PhD, Principal Investigator — University of Michigan
Locations (1):
- Chronic Pain and Fatigue Research Center, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No